CLINICAL TRIAL: NCT07391943
Title: Efficacy of a Self-Guided Cognitive Behavioral Therapy Protocol Via Mobile Application in Patients With Treatment-Resistant Panic Disorder: An Open-Label Trial
Brief Title: Self-Guided CBT Mobile App for Treatment-Resistant Panic Disorder (CBT) Cognitive Behavioral Therapy
Acronym: (CBT)
Status: Completed | Type: Observational
Sponsor: Universidade Federal do Rio de Janeiro (Other)
Responsible Party: Principal Investigator, Luisa Pelucio Ribeiro Barbosa, Researcher, Universidade Federal do Rio de Janeiro
Other Study IDs: UFRJ-2025-002
Record Dates: First submitted 2025-08-16; First posted 2026-02-06 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2025-05

CONDITIONS: Panic Disorder
Keywords: Panic disorder;; Cognitive behavioral therapy;; Mobile application;; Digital intervention;; Self-guided treatment;; Treatment-resistant panic disorder
MeSH Terms: conditions — Panic Disorder

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 8 Weeks
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: Experimental - Self-Guided CBT Mobile App — Eight-session manualized CBT protocol delivered via mobile app, including psychoeducation, cognitive restructuring, relaxation, behavioral activation, assertiveness, and life reorganization, with avatar interface to enhance engagement.

SUMMARY:
Treatment-resistant panic disorder (TRPD) is characterized by persistent panic symptoms despite adequate pharmacological and/or psychotherapeutic treatment. This open-label study is designed to evaluate a self-guided cognitive behavioral therapy (CBT) protocol delivered via a mobile application for adults with TRPD. The intervention consists of eight weekly sessions covering psychoeducation, panic cycle interruption, cognitive restructuring, relaxation techniques, assertiveness training, behavioral strategies, and life reorganization. An avatar is incorporated to enhance engagement and simulate therapeutic presence. Participants continue their usual psychiatric follow-up and pharmacological treatment throughout the study. Outcomes are assessed at baseline and after completion of the intervention using validated measures of panic severity, anxiety, depression, mindfulness, coping strategies, quality of life, and affect.

DETAILED DESCRIPTION:
Panic disorder (PD) is a prevalent anxiety disorder associated with significant functional impairment. Although pharmacotherapy and cognitive behavioral therapy (CBT) are considered first-line treatments, a substantial proportion of patients continue to experience clinically relevant symptoms, characterizing treatment-resistant panic disorder (TRPD). Digital mental health interventions, particularly self-guided CBT delivered via mobile applications, represent a scalable approach to expanding access to evidence-based care.

This open-label study employs an eight-session self-guided CBT protocol delivered through a mobile application for adults diagnosed with TRPD. The intervention is structured into weekly modules addressing psychoeducation about panic disorder, identification and modification of maladaptive cognitions, interruption of the panic cycle, relaxation techniques, assertiveness training, behavioral strategies, and life reorganization. An interactive avatar is included to simulate therapeutic presence and support user engagement.

Participants are recruited from a specialized outpatient clinic and are required to maintain ongoing psychiatric follow-up and stable pharmacological treatment during the study period. Study assessments are conducted at baseline and at the end of the eight-week intervention. Outcome measures include validated self-report instruments assessing panic severity, anxiety symptoms, depressive symptoms, mindfulness, coping strategies, quality of life, and positive and negative affect

ELIGIBILITY:
Inclusion Criteria:

* Age 18-60
* DSM-5 diagnosis of TRPD confirmed by psychiatrist
* Ongoing psychiatric follow-up
* Current pharmacological treatment for PD
* Ability to use smartphone/app

Exclusion Criteria:

* No PD diagnosis
* Other primary psychiatric disorder
* Severe cognitive impairment
* Inability to use the app

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Patients in the panic and respiratory of the Federal University of Rio de Janeiro
Sampling Method: Probability Sample
Enrollment: 45 (Actual)
Dates: Start 2024-11-01 (Actual); Primary Completion 2025-05-30 (Actual); Study Completion 2025-05-30 (Actual)

PRIMARY OUTCOMES:
Beck Anxiety Inventory (BAI) Total Score | Baseline (Week 1) and Post-intervention (Week 8)
  The Beck Anxiety Inventory (BAI) is a 21-item self-report questionnaire designed to assess the severity of anxiety symptoms. Total scores range from 0 to 63, with higher scores indicating greater anxiety severity. The BAI is administered to all participants at baseline and at the end of the intervention.
  Unit of Measure: Points on a scale (0-63)

SECONDARY OUTCOMES:
Beck Depression Inventory-II (BDI-II) Total Score | Baseline (Week 1) and Post-intervention (Week 8)
  The Beck Depression Inventory-II (BDI-II) is a 21-item self-report instrument used to assess the severity of depressive symptoms. Total scores range from 0 to 63, with higher scores indicating greater depression severity. The BDI-II is administered to all participants at baseline and at the end of the intervention.
  Unit of Measure: Points on a scale (0-63)

OTHER OUTCOMES:
Mindful Attention Awareness Scale (MAAS) Total Score | Baseline (Week 1) and Post-intervention (Week 8)
  The Mindful Attention Awareness Scale (MAAS) is a 15-item self-report questionnaire that assesses dispositional mindfulness in daily life. Total scores range from 15 to 90, with higher scores indicating greater mindfulness. The MAAS is administered to all participants at baseline and at the end of the intervention.
  Unit of Measure: Points on a scale (15-90)
WHOQOL-BREF Physical Health Domain Score | Baseline (Week 1) and Post-intervention (Week 8)
  The World Health Organization Quality of Life-BREF (WHOQOL-BREF) Physical Health domain assesses physical aspects of quality of life, including energy, mobility, and daily activities. Domain scores range from 4 to 20, with higher scores indicating better perceived physical quality of life. The domain score is assessed at baseline and at the end of the intervention.
  Unit of Measure: Points on a scale (4-20)
WHOQOL-BREF Social Relationships Domain Score | Baseline (Week 1) and Post-intervention (Week 8)
  The WHOQOL-BREF Social Relationships domain evaluates interpersonal relationships, social support, and personal relationships. Domain scores range from 4 to 20, with higher scores indicating better social quality of life. The domain score is assessed at baseline and at the end of the intervention.
  Unit of Measure: Points on a scale (4-20)
WHOQOL-BREF Environment Domain Score | Baseline (Week 1) and Post-intervention (Week 8)
  The WHOQOL-BREF Environment domain assesses perceptions of safety, home environment, financial resources, access to health care, and opportunities for leisure. Domain scores range from 4 to 20, with higher scores indicating better environmental quality of life. The domain score is assessed at baseline and at the end of the intervention.
  Unit of Measure: Points on a scale (4-20)
Panic and Agoraphobia Scale (PAS) Total Score | Baseline (Week 1) and Post-intervention (Week 8)
  The Panic and Agoraphobia Scale (PAS) is a clinician-administered instrument consisting of 13 items that assess the severity of panic and agoraphobia symptoms. Total scores range from 0 to 52, with higher scores indicating greater symptom severity. The PAS is administered at baseline and at the end of the intervention.
  Unit of Measure: Points on a scale (0-52)

CONTACTS AND LOCATIONS:
Overall Officials: Luisa Pelucio, Dr, Principal Investigator — Universidade Federal do Rio de Janeiro
Locations (1):
- Luisa, Rio de Janeiro, Rio de Janeiro, Brazil

IPD SHARING:
Plan to Share IPD: Yes
Study Protocol
Supporting Information: Study Protocol
Time Frame: For free time
Access Criteria: Just ask for contact information we share.

REFERENCES:
- [Result] Planert J, Machulska A, Hildebrand AS, Roesmann K, Otto E, Klucken T. Self-guided digital treatment with virtual reality for panic disorder and agoraphobia: a study protocol for a randomized controlled trial. Trials. 2022 May 21;23(1):426. doi: 10.1186/s13063-022-06366-x. PMID 35597959
- [Result] Pauley D, Cuijpers P, Papola D, Miguel C, Karyotaki E. Two decades of digital interventions for anxiety disorders: a systematic review and meta-analysis of treatment effectiveness. Psychol Med. 2023 Jan;53(2):567-579. doi: 10.1017/S0033291721001999. Epub 2021 May 28. PMID 34047264
- [Result] Jung HW, Jang KW, Nam S, Kim A, Lee J, Ahn ME, Lee SK, Kim YJ, Shin JK, Roh D. Digital Cognitive Behavioral Therapy for Panic Disorder and Agoraphobia: A Meta-Analytic Review of Clinical Components to Maximize Efficacy. J Clin Med. 2025 Mar 6;14(5):1771. doi: 10.3390/jcm14051771. PMID 40095899
- [Result] Modesto-Lowe V, Adams S, Rossi A. Smartphone Applications: Therapy at Your Fingertips. Prim Care Companion CNS Disord. 2024 Aug 20;26(4):24lr03754. doi: 10.4088/PCC.24lr03754. No abstract available. PMID 39178019
- [Result] Olthuis JV, Watt MC, Bailey K, Hayden JA, Stewart SH. Therapist-supported Internet cognitive behavioural therapy for anxiety disorders in adults. Cochrane Database Syst Rev. 2016 Mar 12;3(3):CD011565. doi: 10.1002/14651858.CD011565.pub2. PMID 26968204
- [Result] Watson D, Clark LA, Tellegen A. Development and validation of brief measures of positive and negative affect: the PANAS scales. J Pers Soc Psychol. 1988 Jun;54(6):1063-70. doi: 10.1037//0022-3514.54.6.1063. PMID 3397865
- [Result] Beck AT, Epstein N, Brown G, Steer RA. An inventory for measuring clinical anxiety: psychometric properties. J Consult Clin Psychol. 1988 Dec;56(6):893-7. doi: 10.1037//0022-006x.56.6.893. No abstract available. PMID 3204199
- [Result] Development of the World Health Organization WHOQOL-BREF quality of life assessment. The WHOQOL Group. Psychol Med. 1998 May;28(3):551-8. doi: 10.1017/s0033291798006667. PMID 9626712
- [Result] Kocalevent RD, Zenger M, Hinz A, Klapp B, Brahler E. Resilient coping in the general population: standardization of the brief resilient coping scale (BRCS). Health Qual Life Outcomes. 2017 Dec 28;15(1):251. doi: 10.1186/s12955-017-0822-6. PMID 29282066
- [Result] Brown KW, Ryan RM. The benefits of being present: mindfulness and its role in psychological well-being. J Pers Soc Psychol. 2003 Apr;84(4):822-48. doi: 10.1037/0022-3514.84.4.822. PMID 12703651
- [Result] Rus-Calafell M, Ehrbar N, Ward T, Edwards C, Huckvale M, Walke J, Garety P, Craig T. Participants' experiences of AVATAR therapy for distressing voices: a thematic qualitative evaluation. BMC Psychiatry. 2022 May 24;22(1):356. doi: 10.1186/s12888-022-04010-1. PMID 35610590
- [Result] Jang B, Yuh C, Lee H, Shin YB, Lee HJ, Kang EK, Heo J, Cho CH. Exploring User Experience and the Therapeutic Relationship of Short-Term Avatar-Based Psychotherapy: Qualitative Pilot Study. JMIR Hum Factors. 2025 Feb 5;12:e66158. doi: 10.2196/66158. PMID 39924261
- [Result] Pagliari C, Burton C, McKinstry B, Szentatotai A, David D, Serrano Blanco A, Ferrini L, Albertini S, Castro JC, Estevez S, Wolters M. Psychosocial implications of avatar use in supporting therapy for depression. Stud Health Technol Inform. 2012;181:329-33. PMID 22954882
- [Result] Pelucio L, Quagliato LA, Cardoso A, Horato N, Nardi AE. Could the use of web-based applications assist in neuropsychiatric treatment? An umbrella review. BMC Psychol. 2025 Mar 26;13(1):302. doi: 10.1186/s40359-024-02263-x. PMID 40140888
- [Result] Pelucio L, Quagliato LA, Nardi AE. Therapist-Guided Versus Self-Guided Cognitive-Behavioral Therapy: A Systematic Review. Prim Care Companion CNS Disord. 2024 Mar 21;26(2):23r03566. doi: 10.4088/PCC.23r03566. PMID 38512281
- [Result] Firth J, Torous J, Nicholas J, Carney R, Pratap A, Rosenbaum S, Sarris J. The efficacy of smartphone-based mental health interventions for depressive symptoms: a meta-analysis of randomized controlled trials. World Psychiatry. 2017 Oct;16(3):287-298. doi: 10.1002/wps.20472. PMID 28941113
- [Result] Pasarelu CR, Andersson G, Bergman Nordgren L, Dobrean A. Internet-delivered transdiagnostic and tailored cognitive behavioral therapy for anxiety and depression: a systematic review and meta-analysis of randomized controlled trials. Cogn Behav Ther. 2017 Jan;46(1):1-28. doi: 10.1080/16506073.2016.1231219. Epub 2016 Oct 7. PMID 27712544
- [Result] Bystritsky A. Treatment-resistant anxiety disorders. Mol Psychiatry. 2006 Sep;11(9):805-14. doi: 10.1038/sj.mp.4001852. Epub 2006 Jul 18. PMID 16847460